CLINICAL TRIAL: NCT07321574
Title: An Open-Label, Multi-Cohort Phase IIb Clinical Study Evaluating the Efficacy and Safety of ABP1011T Tablets in Patients With Advanced Solid Tumors
Brief Title: A Study Evaluating the Efficacy and Safety of ABP1011T Tablets in Patients With Advanced Solid Tumors
Acronym: ABP1011T-03
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai AB PharmaTech Ltd. (Industry)
Collaborators: GCP ClinPlus Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABP1011T-II-03; IND161926 (Other: FDA)
Record Dates: First submitted 2025-11-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: SCLC, Extensive Stage; Advanced Solid Tumors
Keywords: SLCL; Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Based on safety and efficacy data from the prior Phase I/IIa clinical trial (Protocol Number: ABP1011T-I/II-01), priority enrollment is given to participants with advanced solid tumors including small cell lung cancer, esophageal cancer, cervical cancer, bladder cancer, and renal cell carcinoma (excluding osteosarcoma). Cohort A (Cohort A1, Cohort A2, Cohort A3) comprises the small cell lung cancer cohort: Participants must have failed at least two prior systemic therapies. Cohort B enrolls participants with other advanced solid tumors (excluding osteosarcoma).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABP1011T Tablets in Patients with Advanced Solid Tumor (Experimental)
  Interventions: Drug: ABP1011T

INTERVENTIONS:
Drug: ABP1011T — ABP1011T tablets are administered as continuous therapy in clinical studies, with a 21-day treatment cycle. Participants take one tablet orally once daily on an empty stomach (with water, avoiding food for at least 1 hour before and after each dose).

SUMMARY:
This study is a multicenter, open-label, multi-cohort investigation exploring the efficacy and safety of ABP1011T tablets in participants with specific target solid tumors, providing a foundation for subsequent clinical research.

Based on safety and efficacy data from the prior Phase I/IIa clinical trial (Protocol Number: ABP1011T-I/II-01), priority enrollment is given to participants with advanced solid tumors including small cell lung cancer, esophageal cancer, cervical cancer, bladder cancer, and renal cell carcinoma (excluding osteosarcoma). Cohort A (Cohort A1, Cohort A2, Cohort A3) comprises the small cell lung cancer cohort: Participants must have failed at least two prior systemic therapies. Cohort B enrolls participants with other advanced solid tumors (excluding osteosarcoma).

ABP1011T tablets are administered as continuous therapy in clinical studies, with a 21-day treatment cycle. Participants take one tablet orally once daily on an empty stomach (with water, avoiding food for at least 1 hour before and after each dose).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with protocol requirements;
2. Age 18 <= age <= 75 years, male or female;
3. Expected survival >= 12 weeks;
4. ECOG performance status <= 1 point;
5. Patients with advanced solid tumors who have experienced disease progression on standard therapy, intolerance to standard therapy, or lack of effective standard therapy, with histopathological or cytopathological confirmation (priority enrollment for small cell lung cancer, esophageal cancer, cervical cancer, bladder cancer, renal cell carcinoma, or other potentially sensitive tumor types. Cohort A is the small cell lung cancer cohort: includes patients who have failed at least two prior systemic therapies; Cohort B includes patients with other advanced solid tumors); At least one measurable lesion meeting RECIST v1.1 criteria;
6. Recovery from toxic effects of the last prior treatment (CTCAE <= Grade 1, except for specific conditions such as "alopecia" or "hyperpigmentation"), and the investigator determines that the corresponding AE poses no safety risk;
7. Systolic blood pressure <= 140 mmHg, diastolic blood pressure <= 90 mmHg, with no changes in antihypertensive medications or dosages within 7 days prior to the first dose.
8. Organ and bone marrow function levels must meet the following requirements: Bone marrow: Absolute neutrophil count (ANC) >= 1.5 × 10^9/L, platelet count >= 75 × 10^9/L, Hemoglobin >=90 g/L, with no transfusion of platelets or red blood cells within 14 days prior to the first dose, and no transfusion or treatment with biological response modifiers (e.g., granulocyte colony-stimulating factor, erythropoietin, interleukin-11) within 14 days prior to the first dose; Liver function: No history of liver cirrhosis (decompensated cirrhosis Child-Pugh B or C). For patients without liver metastases: serum total bilirubin (TBIL) <= 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 × ULN. Patients with liver metastases must have TBIL <= 2.5×ULN, ALT and AST <= 5×ULN. Renal function: Serum creatinine <= 1.5×ULN, or creatinine clearance > 60 mL/min (Cockcroft-Gault formula); Urine protein qualitative <= 1+; If urine protein qualitative >= 2+, 24-hour urine protein quantification is required. The investigator will determine eligibility based on test results. Coagulation function: Prothrombin time (PT) <= 1.5 × ULN; International Normalized Ratio (INR) <= 1.5 × ULN, and activated partial thromboplastin time (APTT) <= 1.5 × ULN.
9. Female subjects of childbearing potential must undergo a serum pregnancy test within 3 days prior to initiating study medication, with negative results, and must agree to use a medically approved highly effective contraceptive method (e.g., intrauterine device, oral contraceptive, or condom) during the study period and for 6 months after the last study dose. Male subjects with female partners of childbearing potential must agree to use effective contraception during the study period and for 6 months after the last study dose.

Exclusion Criteria:

1. History of or current presence of other malignant tumors, except for the following:

1) Completely resected basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical carcinoma in situ; 2) Completely resected secondary primary cancer with no recurrence within five years; 2. Patients with known hypersensitivity to any component of the study drug or similar agents, or with a history of severe allergic reactions; 3. Patients who have received any of the following treatments or medications prior to the first study treatment: 1) Major surgery or severe trauma within 4 weeks before the first study drug administration (Major surgery is defined as any invasive procedure involving extensive excision or breaching of the mesothelial barrier, such as the pleural cavity, peritoneum, or meninges. However, diagnostic tissue biopsies are permitted). Severe trauma refers to unhealed wounds, ulcers, or fractures; 2) Received Chinese herbal medicine or traditional Chinese medicine for antitumor indications within 2 weeks prior to the first study drug dose.

3) Received antitumor therapy (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, biologic therapy, or tumor embolization) within 4 weeks prior to the first study drug dose; For oral fluoropyrimidine drugs and endocrine therapy, discontinuation <= 2 weeks or 5 half-lives; for nitrosoureas and mitomycin, discontinuation <= 6 weeks. If washout time is inadequate due to scheduling or drug PK characteristics, discussion with the sponsor is required; 4) Wthin 1 week prior to first dose, received potent CYP3A4 or CYP2C9 inhibitors or inducers; 5) Within 1 week prior to first dose, received drugs known to significantly prolong the QT interval (e.g., Class Ia and Class III antiarrhythmics); 6) Concurrent use of antiplatelet agents or anticoagulants during the screening period that cannot be discontinued; 4. Patients with known brain metastases, brainstem metastases, spinal cord metastases, and/or compression, or unstable central nervous system metastases. (However, the following situations may be determined through discussion between the investigator and sponsor: If asymptomatic, or with stable brain metastasis symptoms, and if steroids, anticonvulsants, or mannitol therapy has not been used or has been discontinued for >=4 weeks prior to the first study dose, and the investigator determines the benefits outweigh the risks, the subject may be considered for screening and enrollment); 5. Patients with symptomatic, disseminated visceral disease at an advanced stage who are at risk of life-threatening complications in the short term, or patients with pleural effusion, ascites, or pericardial effusion who underwent paracentesis or thoracentesis within three weeks prior to the first study dose; 6. Patients with imaging evidence of tumor encasement or infiltration of major vessels (e.g., pulmonary artery, pulmonary vein, superior vena cava, inferior vena cava), or significant tumor invasion into adjacent organs (aorta, trachea, gastrointestinal tract) adjacent to esophageal or gastrointestinal lesions, resulting in high risk of hemorrhage or fistula formation; and patients who have undergone tracheal stent placement.

7. Within 6 months prior to screening, presence of cardiovascular disease meeting any of the following criteria: 1) Congestive heart failure with cardiac function >= New York Heart Association (NYHA) Class II; left ventricular ejection fraction (LVEF) < 50%; 2) Severe arrhythmia requiring medication; 3) QTcF (Fridericia formula) > 450 msec in males or > 470 msec in females, or presence of risk factors for torsades de pointes, such as clinically significant hypokalemia as determined by the investigator, history of familial long QT syndrome, or familial arrhythmia history (e.g., Wolff-Parkinson-White syndrome); and abnormal troponin levels; 4) Myocardial infarction, severe/unstable angina, cardiac revascularization, cerebrovascular accident, or similar events within six months prior to dosing; 5) History of >= Grade 3 thromboembolic events within the past 2 years, or currently receiving thrombolytic or anticoagulant therapy due to high thrombotic risk; 8. Electrolite disturbances during screening; 9. Uncontrolled systemic diseases despite treatment, such as diabetes; 10. Current acute pulmonary disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute pulmonary disease, or treatable reflex interstitial pneumonia; 11. Patients with a clear tendency toward gastrointestinal bleeding, including the following conditions: presence of locally active ulcerative lesions with fecal occult blood test (>=2+); history of melena or hematemesis within the past 2 months; patients deemed by the investigator to be at risk for major gastrointestinal hemorrhage; 12. History of or current unhealed gastrointestinal perforation or visceral fistula; 13. Evidence of active infection:

1. Hepatitis B (HBV) (requiring both positive hepatitis B surface antigen (HBsAg) and HBV-DNA levels exceeding the center's specified detection limit);
2. Hepatitis C (requiring both HCV antibody [HCV-Ab] positivity and HCV-RNA levels exceeding the lower limit of detection for the analytical method);
3. Active local or systemic infection requiring systemic antimicrobial therapy within 4 weeks prior to first dosing, or unexplained fever >38.5°C during screening/prior to first dosing;
4. Active pulmonary tuberculosis infection identified through medical history or CT examination, or history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or history of active pulmonary tuberculosis infection more than 1 year prior without formal treatment; 14. Individuals with positive human immunodeficiency virus (HIV RNA) or Treponema pallidum antibody status; 15. Presence of multiple factors affecting oral medication administration (e.g., inability to swallow, chronic diarrhea, intestinal obstruction), or conditions judged by the investigator to severely impair gastrointestinal absorption; 16. History of confirmed neurological or psychiatric disorders, including epilepsy, dementia, depression, etc.; 17. Patients with alcohol or drug dependence, a history of needle phobia or blood phobia, or inability to tolerate venous blood collection; 18. Habitual consumption of grapefruit juice or excessive amounts of tea, coffee, and/or caffeinated beverages, with inability to discontinue during the trial period; 19. Received any investigational drug within 4 weeks prior to first dosing, or concurrent participation in another clinical study (except: participation in an observational, non-interventional clinical study; being in the follow-up period of an interventional clinical study; or completion of the previous study drug administration more than 5 half-lives ago); 20. Female patients who are pregnant or breastfeeding; 21. Patients deemed unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-11-28 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Relief (DOR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Sustained Response Rate | Up to approximately 2 years
  Proportion of subjects with DoR ≥ 6 months after first dose (based on RECIST v1.1).
Overall Survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.
Two-Year Overall Survival Rate | Up to approximately 2 years
  Two-Year Overall Survival Rate
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to approximately 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaocheng Second People's Hospital, Liaocheng, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Neijiang First People's Hospital, Neijiang, Sichuan
  - Shanghai East Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or any presentations.
Time Frame: After the trial completed.
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.